CLINICAL TRIAL: NCT04052022
Title: Paradoxical Tuberculosis Reactions in Patients Without HIV Infection
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190133; 19-I-0133
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-26

CONDITIONS: Tuberculosis
Keywords: Auto-Antibody Production; Host Genetic Predisposition; Immune Reconstitution Inflammatory Syndrome; Biomarkers; Pathogenesis; Natural History
MeSH Terms: conditions — Tuberculosis; Immune Reconstitution Inflammatory Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with TB who have already initiated treatment and are suspected to have paradoxical reactions
- 2: Patients with TB who have already initiated treatment without signs of paradoxical reactions (control)

SUMMARY:
Background:

Most people with tuberculosis (TB) feel better after starting treatment. But for some people, the opposite happens. They may feel better at first, but then suddenly get worse. This is a paradoxical reaction. Researchers want to better understand what causes this reaction and what happens after someone has it.

Objective:

To learn about paradoxical reactions to TB treatment.

Eligibility:

Adults 18 and older diagnosed with confirmed or suspected TB and currently on treatment for at least 2 weeks, with or without signs/symptoms of a paradoxical inflammatory reaction.

Design:

Participants will be screened with a physical exam and medical history. They will give blood and urine samples.

Eligible participants will visit either the NIH Clinical Center or the Mexico Clinic sites 3 times over 6 to 18 months. Each visit will take 7 hours to complete; visits may be scheduled over more than 1 day. Participants may have more visits if their TB symptoms change.

Participants will give blood, urine, and sputum samples. They will have adverse event assessments. They will have 2 to 3 positron emission tomography/computed tomography (PET/CT) scans. PET/CT scans make pictures of the inside of the body. For this, participants will lie on a table that slides into a donut-shaped scanner. They will get a small amount of radioactive dye through an IV, which is a small plastic tube placed in a vein in the arm using a needle.

Participants may have optional apheresis at the NIH site only. For this, blood is taken from a needle in one arm. White blood cells are separated from the rest of the blood. The rest of the blood is returned through a needle in the other arm.

DETAILED DESCRIPTION:
Paradoxical reaction in non-HIV tuberculosis (TB) is a clinical and/or radiologic worsening of a patient s pre-existing TB while receiving anti-TB medications. This phenomenon has been clinically well described for many years and is thought to occur in 10%-25% of HIV-negative patients starting treatment for TB. Paradoxical reactions are diagnosed by excluding other possible causes for worsening of TB signs and symptoms, such as a second infection or treatment failure. However, challenges in culturing TB can complicate early diagnosis of paradoxical reactions.

This is a multisite, international observational study intended to improve understanding of the pathogenesis of paradoxical response to treatment in TB-infected patients who do not have HIV. Each site will follow up to 20 patients with TB who have already initiated or have previously completed treatment and are suspected to have paradoxical reactions, as well as about 40 patients taking TB treatment without signs of paradoxical reactions (controls). All participants will have regular study visits for clinical assessments, blood and sputum collections, positron emission tomography-computed tomography (PET/CT) scans, and optional leukapheresis. Radiography and laboratory evaluations will be performed to identify biomarkers, clinical signs, and molecular explanations for paradoxical reactions. Better understanding of characteristics of paradoxical reactions will assist in earlier diagnosis or even prediction.

ELIGIBILITY:
* INCLUSION CRITERIA:

Suspected Paradoxical Reaction Group Criteria:

1. Aged greater than or equal to 18 years.
2. Diagnosed with confirmed (microbiologically or with molecular methods) or suspected (clinical plus or minus histologic diagnosis) TB and currently on ATT for a minimum of 2 weeks, or have completed ATT, with at least 2 of the following signs/symptoms of a paradoxical inflammatory reaction:

   * Recrudescent symptoms of TB after initial clinical improvement.
   * Change in physical exam after initial clinical improvement suggestive of new inflammatory process (e.g., lymphadenopathy or new findings on pulmonary exam).
   * Worsening radiographic evidence of disease after initiation of treatment, as compared with imaging prior to or earlier in treatment.
   * Laboratory evidence of acute inflammatory response, including the development of leukocytosis (white blood cell count > 10,000 cells/microL) or a change of C-reactive protein (CRP) > 5 mg/L compared to prior laboratory values.
   * Worsened organ function after initial clinical improvement.
3. The above sign/symptom(s) cannot be explained by a newly acquired infection, clinical course of a previously recognized infectious agent, side effects of the ATT, the presence of drug resistance, or any other condition except for paradoxical reaction.
4. Willingness to allow storage of blood or tissue samples for future research.
5. Ability of participant to understand study requirements and give informed consent.
6. Has a primary care physician and is being followed by the local Department of Health for their TB (or has plans to arrange after enrollment if enrolled early in course from inpatient transfer).

Control Group Criteria:

1. Aged greater than or equal to 18 years.
2. Diagnosed with confirmed (microbiologically or with molecular methods) or suspected (clinical plus or minus histologic diagnosis) TB.
3. Presenting 2 to 4 months after starting ATT to match timing of paradoxical reactions.
4. Willingness to allow storage of blood or tissue samples for future research.
5. Ability of participant to understand study requirements and give informed consent.
6. Has a primary care physician and is being followed by the Department of Health for their TB (or has plans to arrange after enrollment if enrolled early in course from inpatient transfer).

EXCLUSION CRITERIA:

Individuals in either group who meet any of the following criteria will be excluded from study participation:

1. HIV infection. (Individuals with HIV infection may be eligible for a separate study exclusively evaluating persons living with HIV.)
2. Pregnant or breastfeeding.
3. Uncontrolled psychiatric disease, substance use, or inappropriate conduct unsuitable for a research study.
4. Malignancy requiring imminent or ongoing treatment including radiation, chemotherapy, or immunotherapy.
5. Debilitating or chronic conditions that would limit ability to participate in the study.
6. Emergent or urgent clinical conditions not due to studied disease of interest requiring immediate treatment that would be unsuitable for a research study. These patients would be transferred to an emergency room and able to rescreen when condition has been stabilized.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from clinics in the surrounding Washington, DC area for the NIH site; and from clinics in Mexico for the foreign site
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Immunologic and radiographic responses of TB patients with suspected paradoxical reactions. | Throughout study
  Characterize immunologic and radiographic responses of TB patients with suspected paradoxical reactions.

SECONDARY OUTCOMES:
Biomarkers and/or microbiologic burden correlate with paradoxical TB reactions. | Throughout study
  Determine whether biomarkers and/or microbiologic burden correlate with paradoxical TB reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Maura M Manion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Mexican Emerging Infectious Diseases Clinical Research Network (LaRed), Alcaldia Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
No plan at this time.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0133.html